CLINICAL TRIAL: NCT01836770
Title: Epidural Contrast Flow Patterns of Transforaminal Epidural Steroid Injections Using the Inferior-Anterior Position as the Final Needle Tip Position.
Brief Title: Epidural Contrast Flow Patterns of TESI Using the Inferior-Anterior Position as the Final Needle Tip Position.
Status: Terminated | Type: Observational
Why Stopped: lack of enrollment; terminated by the Principal Investigator
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: Kambin
Record Dates: First submitted 2013-01-07; First posted 2013-04-22 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Lumbosacral Radiculopathy; Lumbar Herniated Nucleus Pulposus
Keywords: Transforaminal Epidural Steroid Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transforaminal Epidural Steroid Injection: Patients with a history of lumbosacral radiculopathy or lumbar herniated nucleus pulposus, scheduled for Transforaminal Epidural Steroid Injection.

SUMMARY:
The purpose of this study is to describe the contrast flow patterns in the epidural space using the inferior-anterior approach with continuous fluoroscopic guidance, and determine how well this approach correlates with appropriate contrast flow patterns and with analgesia at follow up. This knowledge may prove useful in guiding physician practice patterns in the non-surgical management of low back pain.

Hypothesis: The investigators hypothesize that there will be suitable (ventral/anterior) epidural contrast spread based on inferior-anterior needle-tip position, particularly with appropriate needle tip position.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* History of lumbosacral radiculopathy or lumbar herniated nucleus pulposus
* Scheduled for TFESI at GW Spine and Pain Center

Exclusion Criteria:

* Pregnant or plan on becoming pregnant
* Have undergone TFESI in the past year
* Opioid habituation
* Lumbo-sacral stenosis
* Lumbar surgery
* Lumbar spondylolisthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: George Washington Spine and Pain Center patients.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2013-06-20 (Actual)

PRIMARY OUTCOMES:
Contrast flow patterns | 3 Months
  Contrast flow patterns will be used as the primary outcome measure. The statistical test to be employed is to compare the proportions of patients in the study who experienced posterior flow, anterior flow and if that anterior flow had spread to more than 1 vertebral level in either direction, what that direction was, and the presence or absence of vascular flow.

SECONDARY OUTCOMES:
VAS pain score | 3 months
  VAS Pain Score - The statistical test to be employed is Wilcoxon Signed Rank Test to compare if there is a difference in pain score at appointments 1 months and 3 months post-injection relative to pre-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Mehul J Desai, MD MPH, Principal Investigator — George Washington Spine and Pain Center
Locations (1):
- George Washington Spine and Pain Center, Washington D.C., District of Columbia, United States